CLINICAL TRIAL: NCT02311764
Title: Single Arm Open Label Phase II Pilot Study of Carboplatin in Patients With Metastatic Castrationresistant Prostate Cancer (CRPC) and PTEN Loss and/or DNA Repair Defects
Brief Title: Carboplatin in Castration-resistant Prostate Cancer
Acronym: PRO-PLAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Aurelius Omlin (Other)
Collaborators: Teva Pharma (Industry); University Hospital, Zürich (Other)
Responsible Party: Sponsor-Investigator, Aurelius Omlin, MD, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTU-14005
Record Dates: First submitted 2014-12-02; First posted 2014-12-08 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin (Experimental): Carboplatin will be administered weekly
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be administered weekly

SUMMARY:
Open label, non-randomised phase II clinical pilot study

DETAILED DESCRIPTION:
Pilot Study of weekly Carboplatin in Patients with Advanced Metastatic Castration-Resistant Prostate Cancer (CRPC) and DNA repair defects

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent
2. Adult patients with histological diagnosis of adenocarcinoma of the prostate.
3. Metastatic Castration-Resistant Prostate Cancer (mCRPC)
4. Progression after at least one taxane-based chemotherapy (or contraindication against taxanes) and at least one therapy with a newer hormonal agent (Cyp17 inhibitor or a new generation AA like enzalutamide).
5. DNA repair defects as per central assessment
6. Eastern Cooperative Oncology Group (ECOG) performance Status (PS) 0 - 2
7. Progression of disease by any of the criteria listed here:

   * PSA utilizing PCWG 2 criteria
   * Bone scan
   * RECIST 1.1
8. Adequate organ and bone marrow function as evidenced by:

   * Haemoglobin ≥8.0 g/dL
   * Absolute neutrophil count ≥1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * AST and/or ALT < 2.5 x ULN, in the presence of liver metastases: AST ≥5 x ULN, ALT <5 x ULN
   * Total bilirubin < 2.0 x ULN (except for patients with Gilbert's disease)
   * Creatinine Clearance ≥30ml/min
9. Patient must agree in the biomarker studies including the fresh tumour biopsies

Exclusion Criteria:

1. Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product Carboplatin
2. Prior treatment with any prior platinum based chemotherapy,
3. Major surgery within 4 weeks prior to planned start of treatment
4. Known brain or leptomeningeal involvement unless clinically stable and on stable dose of steroids
5. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
6. Previous enrolment into the current study
7. Active secondary malignancy that requires systemic therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Response | Time Frame: Up to the end of the treatment phase (ie, approximately 6 months
  Soft tissue or PSA Response

SECONDARY OUTCOMES:
Rate of PSA declines of ≥30% | Time Frame: At 12 weeks and up to the end of the treatment phase (ie, approximately 6 months)
  PSA
OS | Time Frame: livelong follow-up
  Overall survival (OS) form start of Carboplatin
rPFS | Time Frame: Up to the end of the treatment phase (ie, approximately 6 months
  Radiological progression-free survival (rPFS) from start of carboplatin
PSA | on studyTime Frame: Up to the end of the treatment phase (ie, approximately 6 months
  Time to PSA progression
Safety as per CTC AEv4.03 | on studyTime Frame: Up to the end of the treatment phase (ie, approximately 6 months
  Number of patients with adverse events
Disease control rate | On studyTime Frame: Up to the end of the treatment phase (ie, approximately 6 months
  Disease control rate at 12 and 24 weeks (defined as SD, PR, CR, see response criteria
PTEN loss | Pre-study biopsy sample
  Evaluation of PTEN loss by FISH (Frequency and correlation with IHC)

CONTACTS AND LOCATIONS:
Overall Officials: Aurelius G Omlin, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (3):
- Switzerland (3):
  - Cantonal Hospital Chur, Chur, Kanton Graubünden
  - Luzern Cantonal Hospital, Lucerne
  - Cantonal Hospital St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Undecided